# Statistical Analysis Plan

An open-label, randomized, single-dose, parallel group study to investigate the pharmacokinetics of oxycodone and naloxone from oxycodone/naloxone (OXN) prolonged release (PR) tablet 5/2.5 mg (OXN 5/2.5)and20/10 mg (OXN 20/10) in Chinese patients with moderate to severe chronic non-malignant pain.

Product Name: Oxycodone Naloxone Prolonged Release Tablets (OXN PR)

Sponsor: Mundipharma (China) Pharmaceutical Co., Ltd.

Version 1.0: Mar 1, 2017

#### STATISTICAL ANALYSIS PLAN

Study title: An open-label, randomized, single-dose, parallel group study to

investigate the pharmacokinetics of oxycodone and naloxone from oxycodone/naloxone (OXN) prolonged release (PR) tablet 5/2.5 mg (OXN 5/2.5)and20/10 mg (OXN 20/10) in Chinese patients with

moderate to severe chronic non-malignant pain.

**Sponsor:** Mundipharma (China) Pharmaceutical Co., Ltd.

**Investigator:** Professor Hu Bei, Peking Union Medical College Hospital

Professor Zeng Xiao-feng, Peking Union Medical College Hospital

Study doctor: Dr. Chen Xia, Peking Union Medical College Hospital

Clinical trial

2011L01178,2011L01179,2012L02501,2012L02502

approval number:

**Protocol number:** OXN08-CN-101

**Sponsor:** 18F, Building D, CITC, A6 Jianguomenwai Street,

Chaoyang District, Beijing, P. R. China

Postal Code: 100022

Telephone: +861065636800 Fax: +8610 65636700

**Version/Date:** 1.0: Mar 1, 2017

#### **Confidentiality Statement**

The information contained in this document, the unpublished data in particular, is owned or controlled by Mundipharma (China) Pharmaceutical Co., Ltd. The information is hereby made available in a confidential form to you as an investigator, a potential investigator or a consultant for reviews by you, your staffs and relevant ethics committee. All information should only be used in clinical study of the test drug you are authorized to carry out as described in this protocol. Except for the necessity to disclose certain information to the possible subject to certain extent when obtaining the informed consent, the information shall not be disclosed to any third parties without written permission of Mundipharma (China) Pharmaceutical Co., Ltd.

## **Table of Contents**

| STATISTICAL ANALYSIS PLAN | 2 |
|-------------------------------------------|----|
| Signature page | 1 |
| Table of abbreviations | 3 |
| 1. Overview | 4 |
| 1.1 Study Rationale | 4 |
| 1.2 Study objectives | 4 |
| 1.3 Study design | 5 |
| 1.3.1 Study design | 5 |
| 1.3.2 Determination of sample size | 6 |
| 1.3.3 Blinding | 6 |
| 1.4 Guidelines | 6 |
| 2. Study subjects | 6 |
| 2.1 Subject arrangement | 6 |
| 2.2 Analytical sets | 6 |
| 2.3 Protocol deviation | 7 |
| 2.4 Demographics and baseline analysis | 7 |
| 2.4.1 Demographics | 7 |
| 2.4.2 Concomitant Medication | 7 |
| 2.5 Determination of treatment compliance | 7 |
| 3. Pharmacokinetic evaluation | 7 |
| 3.1 Analytical data | 7 |
| 3.2 Pharmacokinetic evaluation | 7 |
| 3.2.1 Calculation of PK parameter | 7 |
| 3.2.2 Evaluation of dose-proportionality | 9 |
| 3.3.3 Data handling conventions | 10 |
| 4. Safety assessment | 11 |
| 4.1 Analytical data | 11 |
| 4.2 Exposure data | 11 |
| 4.3 Adverse events | 11 |
| 4.3.1 Serious adverse events | 11 |
| 4.4 Evaluation of laboratory tests | 11 |
| 4.5 Vital signs | 12 |
| 4.6 Physical examination | 12 |
| 4.7 ECG evaluation | 12 |
| 4.8 Evaluation of pain scores | 12 |
| 5. Quality control | 12 |
| 6. List of Tables. | 13 |
| 6.1 List of Tables. | 13 |
| 6.2 List of figures | 13 |
| 6.3 Table of listings | 14 |
| 7. References | 14 |
| 8. Examples of tables | 15 |
| Tables | 15 |

| Figures | 24 |
|---------|----|
| Listing | 25 |

| CI. | 4 | |
|------|-------|------|
| Sign | ature | nage |
| ~-5 | | P 5 |

| Writer Statistician Yiwen Wu Clinical Pharmacology Research Center of Peking Union Medical College Hospital | |
|---|---|
| Signature | Date |
| Reviewer Sub-investigator Xia Chen, Associate Professor Clinical Pharmacology Research Center of Peking Union Medical College Hospital | |
| Signature | Date |
| Reviewer Bioanalysis investigator Hongyun Wang, Associate Professor Clinical Pharmacology Research Center of Peking Union Medical College Hospital | |
| Signature | Date |

| Reviewer<br>Clinical lead | |
|---|---|
| York Peng | |
| Mundipharma (China) Pharmaceutical Co., Ltd. | |
| Signature | Date |
| Approver | |
| Principle investigator | |
| Pei Hu, Professor | |
| Clinical Pharmacology Research<br>Center of Peking Union Medical<br>College Hospital | |
| Signature Signature | Date |

## **Table of abbreviations**

| Abbreviation | Annotation |
|---|---|
| AE | Adverse events |
| AUC <sub>0-inf</sub> | Area under plasma drug concentration-time curve from zero time to |
| | infinity |
| AUC <sub>0-t</sub> | Area under plasma drug concentration-time curve from zero time to |
| | the last measurement |
| AUC_%Extrap | Percentage of extrapolated area |
| BLQ | Below Limit of Quantification |
| BMI | Body mass index |
| CFDA | China Food and Drug Administration |
| C <sub>max</sub> | Peak plasma concentration |
| CRF | Case report form |
| ECG | Electrocardiogram |
| Lambda_z | Elimination rate constant |
| LLOQ | Lower Limit of Quantification |
| IMP | Investigational medicinal product |
| MedDRA | Medical Dictionary for Regulatory Activities |
| NC | Not calculate |
| ND | Not detectable |
| OXN PR | Oxycodone Naloxone Prolonged Release Tablets |
| PK | Pharmacokinetics |
| SAE | Serious adverse events |
| T <sub>max</sub> | Time to peak plasma concentration |
| t <sub>1/2</sub> | Elimination half-life |

#### 1. Overview

#### 1.1 Study Rationale

Mundipharma Research GmbH & Co. KG and independent affiliates (NPRL and Purdue Pharma L.P) have developed a novel compound prolonged-release analgesic tablet composed of an opioid agonist oxycodone and an opioid antagonist naloxone. Oxycodone is a sustained-release dosage form of opioid analgesics indicated for moderate-severe pain.

Adding naloxone component to the fixed combination can offset opioid-induced constipation by locally blocking the effect of oxycodone on opioid receptors in the intestines. In addition, due to the presence of opioid receptor antagonist naloxone, lower abuse rate is expected with Oxycodone Naloxone Prolonged Release Tablets (OXN PR) than with single-component sustained-release opioids when the tablet is grounded for intravenous or intranasal administration. Opioids are the cornerstone of chronic pain management. It has been shown that opioid sustained-release drugs are effective for pain management; however, the adverse events (AE) have limited the ability to appropriately increase opioid doses to manage the pain. Among patients who receive opioid to manage pain, the induced constipation is a frequently occurring severe adverse event (SAE). Laxatives are the currently recommended treatment, but many patients frequently discontinue opioid therapy because opioid-induced constipation continues to exist with medication. Therefore, it is highly beneficial to minimize the occurrence or reduce the severity of constipation. In the current compound formulation, the high first-pass effect of naloxone is considered to be an advantage: the local action of naloxone in the intestine can improve intestinal function; given the low systemic bioavailability of naloxone, however, the analgesic activity of oxycodone is not inhibited. The results of all clinical studies conducted so far have shown no significant effect on the analgesic efficacy after compound OXN PR formulation is administered, but the patients indeed benefited from relieved constipation and tolerated this product very well.

#### 1.2 Study objectives

The primary objectives of this study are:

- To determine the pharmacokinetic (PK) characteristics of oxycodone, naloxone and its metabolites in Chinese patients (with moderate to severe chronic non-malignant pain).
- To assess, in a single dose investigation, the dose-proportionality of OXN.

#### 1.3 Study design

#### 1.3.1 Study design

This is an open-label, randomized, single-dose and parallel-group study. A total of 24 subjects are expected to be enrolled and randomized at 1:1 ratio into single-dose Oxycodone Naloxone Prolonged Release Tablets (OXN PR) 5/2.5 mg group or OXN PR 20/10 mg group, each group includes 12 subjects who will orally receive OXN PR active drug. If fewer than 12 subjects in each group have completed this study, more subjects will be included.

Subjects will attend a screening visit within 14days of the first (OXN) dosing day (Day 1).

Eligible subjects will then check into the study unit on the day before OXN dosing (Day -2). Subjects will be administered their OXN dose the next 2 morning (Day 1), following an overnight fast.

There will be 24 subjects with moderate to severe chronic non-malignant pain enrolled in this single-dose study, to be comprised of males and females aged 18-65 years. Blood samples will be collected in tubes containing the anticoagulant EDTA pre-dose and up to 48 hours after administration of OXN. Subjects remain in the study unit up to 48+2 hours after OXN dosing.

Vital signs (pulse, blood pressure, respiration rate) will be monitored pre-dose and then at 1, 2, 4, 6, 8, 12, 24, 36, 48 hours after OXN dosing. Auxiliary temperature will be monitored pre-dose, 24, 36, 48 hours after OXN dosing.

AEs will be recorded throughout the study. Subjects will attend a post-study evaluation 48±2 hours after OXN dosing (in the case of discontinuation from the study).

Figure 1: Study Diagram
Single-dose administration:



Screening period: Day -14 to Day -2

Treatment and sampling period: 2 days

Group A: **OXN PR** 5/2.5 mg, 1 tablet

Group B: OXN PR 20/10 mg, 1 tablet

Post-study evaluation: 1 day

#### 1.3.2 Determination of sample size

No formal sample size calculations will be performed. 24 subjects (12 in each dosage group) are regarded as sufficient according to CFDA regulation requirement. If subject withdraw from the study, subject replacement is needed.

#### 1.3.3 Blinding

Not applicable.

#### 1.4 Guidelines

This statistical plan will follow the SOP of Clinical Pharmacology Research Center of Peking Union Medical College Hospital and the requirements of China authority.

#### 2. Study subjects

#### 2.1 Subject arrangement

The number and percentage of subjects completed and discontinued from this trial should be included in the statistical analysis report; meanwhile, the information of the subjects discontinued from the trial, including the reason for discontinuation, should be listed.

#### 2.2 Analytical sets

#### • Intention-to-treat (ITT) population

ITT population consists of all randomized subjects who meet the inclusion and exclusion criteria.

#### Safety set (SS)

Safety set is a subset of ITT population and consists of all subjects who receive at least 1 dose and have evaluable safety data.

#### • PK analysis set (PKS)

PK analysis set is a subset of ITT population and consists of all subjects who receive at least 1 dose and have evaluable PK data. It should also be noted: according to the protocol, subjects who experience vomiting within 12hr after OXN is administered should not be included in the PKS.

All the above analysis sets will be determined in data review report.

#### 2.3 Protocol deviation

Primary and secondary protocol deviations should be listed in the statistical analysis report. (Note: Major PD will be identified in the data review report.)

#### 2.4 Demographics and baseline analysis

#### 2.4.1 Demographics

Safety set (SS) will be used to summarize and list demographic and baseline variables. Individual demographic and baseline characteristic data should be listed in the statistical analysis report.

Demographic variables such as age, gender, weight, height and ethnicity will be listed by dose group and subject; descriptive statistical analysis will be conducted by dose group. The continuous variables in the table should list the descriptive statistical results, while the categorical variables should list the frequency and percentage.

Medical History should be listed in the statistical analysis report.

#### 2.4.2 Concomitant Medication

The list of Concomitant Medication should include all combined use of drugs in safety sets by drug and drug category.

#### 2.5 Determination of treatment compliance

The beginning date, ending date and time of administration in these subjects will be listed in the statistical analysis report.

#### 3. Pharmacokinetic evaluation

#### 3.1 Analytical data

PK evaluation will be based on the data of all subjects in PKS.

#### 3.2 Pharmacokinetic evaluation

#### 3.2.1 Calculation of PK parameter

If there is no protocol deviation (e.g. failure to take study drug) that may affect PK endpoint variables (e.g. AUC, Cmax) during this trial, the subject will be included in PKS.

Non-compartmental analysis method (Linear Up Log Down) of Phoenix WinNonlin 6.3

(Pharsight Corp., Mountain View, CA, USA) software will be used not only to calculate PK parameters of oxycodone and its metabolites (noroxycodone, oxymorphone and noroxymorphone), and naloxone and its metabolites (6 $\beta$ -naloxol, naloxone-3-glucuronate and 6 $\beta$ -naloxol-3-glucuronate) but also to conduct descriptive statistical analysis, including the following parameters:

| Parameters | Definitions | Calculation methods |
|---|---|---|
| AUC <sub>0-inf</sub> | The area under the plasma concentration-time curve from time 0 to infinity | AUC <sub>0-inf</sub> =AUC <sub>0-t</sub> +(Clast/Lambda_z), where Clast is the corresponding blood concentration at the last measurable time point Tlast. |
| AUC <sub>0-t</sub> | The area under the plasma concentration-time curve from time 0 to the last measurable concentration (Clast) | Linear/ log trapezoidal method |
| Cmax | Maximum plasma concentration | It shall be obtained directly from observation data. |
| Lambda_z | Elimination rate constant [1/ hr] | The elimination rate constant shall be calculated using the linear regression of log-linear concentration-time curve. The time point can be included only if corresponding linearity decreases. |
| T1/2 | Half-life of elimination [hr] | T½=ln(2)/Lambda_z. The time point can be included only if corresponding linearity decreases. |
| Tmax | Time to peak blood concentration [hr] | Time to peak blood concentration present for<br>the first time on the time axis shall be obtained<br>from observation data. |
| AUC_%Extrap | The percentage AUC extrapolated [%] | The percentage of area under the plasma concentration-time curve from the last measurable concentration time point after dosing $t$ to infinity in $AUC_{0-inf}$ |

Descriptive statistical analysis of the PK parameters of oxycodone and its metabolites (noroxycodone, oxymorphone and noroxymorphone), and naloxone and its metabolites (6β-naloxol,

naloxone-3-glucuronate and 6β-naloxol-3-glucuronate) are conducted by dose group. The descriptive statistics include mean, standard deviation, coefficient of variation, minimum and maximum.

The mean concentration-time curve (Mean $\pm$ SD) for oxycodone and its metabolites (noroxycodone, oxymorphone and noroxymorphone), naloxone and its metabolites (6 $\beta$ -naloxol, naloxone-3-glucuronate and 6 $\beta$ -naloxol-3-glucuronate) are plotted by dose group.

#### 3.2.2 Evaluation of dose-proportionality

The linear mixed effect model (treatment as fixed factor, subject as random effect) will be used for exploratory evaluation of the dose-proportionality of for oxycodone, naloxone and metabolites ( $AUC_{0-48h}$ , AUC0-inf and  $C_{max}$ ).

#### **Evaluation objectives**

The objective of drug dose-proportionality assessment is to determine whether there is a proportional relationship between the dose and exposure level of study drug, which is usually evaluated by measuring the relationship between concentration-related PK parameters (e.g.  $AUC_{0-48hr}$ , AUC0-inf and  $C_{max}$ ) and doses.

#### Method for the evaluation of drug dose-proportionality

#### Power Model

Power Model <sup>[1,2]</sup> is used to find the point estimate and 90% confidence interval (CI) for the degree of drug dose-proportionality deviation between the lowest dose and the highest dose during this trial; then, the acceptable range after correction by the dose range (see texts below for correction method) is used to determine whether the drug demonstrates linearity within this dose range. If 90% CI for  $\beta$  falls within ( $\theta_L$ ,  $\theta_U$ ), the drug dose linearly can be established within this dose range; if 90% CI for  $\beta$  partially falls within ( $\theta_L$ ,  $\theta_U$ ), the drug dose linearly cannot be fully established within this dose range, but 90% CI for deviation of the drug dose linearly falls within ( $\beta_L$ ,  $\beta_U$ ).

Correction method of the acceptance range:  $\gamma$ =maximum dose/minimum dose;  $\theta_L = \exp((\beta_L - 1) * \ln \gamma)$ ;  $\theta_U = \exp((\beta_U - 1) * \ln \gamma)$ ;  $\beta_L$  is the lower limit of CI for  $\beta$ ;  $\beta_U$  is the upper of CI for  $\beta$ . The  $\beta$  estimate and its CI are obtained with the mixed model after logarithmic conversion of PK parameters. The  $\beta$  estimate,  $\theta_L$  and  $\theta_U$  should be all listed in statistical analysis report.

#### 3.3.3 Data handling conventions

#### 3.3.3.1 Basic principles of PK data handling

The handling of PK concentration data and the calculation of PK parameters in this trial should comply with following basic principles:

- 1) When calculating PK parameters of data obtained at drug concentration below the lower limit of quantitation (BLQ), the value should be replaced with zero if occurring before  $T_{max}$  and the value should be replaced with ND if the BLQ occurs after  $T_{max}$ ;
- 2) After  $T_{max}$ , if measurable concentration appears after two consecutive NDs, it should be replaced with ND if there is no measurement error;
- 3) When descriptive statistics for concentration at each time point are calculated, all data below LLOQ are not brought into the calculation;
- 4) When descriptive statistics for concentration at each time point are calculated, if more than 1/3 of the individual data is not brought into the calculation, the descriptive statistics at that time point will not be calculated and are represented with NC;
- 5) When the descriptive statistics of concentrations at each time point are calculated, if a subject vomits within 12 hours after the administration, then this subject will not be included in the statistical analysis of PK, but the plasma drug concentration at the corresponding time point will be provided in the listing;
- 6) If the extrapolated area of AUC is greater than 20% of AUC<sub>0-inf</sub>, AUC<sub>0-inf</sub><0.8, then the AUC<sub>0-inf</sub> will neither be included nor be brought into any statistical analysis of AUC<sub>0-inf</sub>;
  - 7) The calculation of all PK parameters employs the actual time and measured concentration.
- 8) All individual plasma drug concentration retains 3 significant digits, while the descriptive statistical results (mean and standard deviation) retain 2 digits after the decimal point; individual PK parameters and their descriptive results retain 2 significant digits.
  - 9) Handling of missing data:

When missing data is determined, the test results corresponding to this point will not be brought into the calculation of relevant statistics.

#### 3.3.3.2 Statistical method for PK analysis

Descriptive statistics of PK parameters include the number of cases (N), arithmetic mean (Mean), standard deviation (SD), coefficient of variation (CV), minimum (Min), median and maximum (Max). The descriptive statistics of PK parameters (mean, standard deviation, coefficient of variation, minimum, median and maximum) will be provided by the listing of test drugs. All statistical analysis will employ SAS® 9.3.

#### 4. Safety assessment

All statistical analysis will employ SAS® 9.3.

#### 4.1 Analytical data

Safety analysis will be based on the data of all subjects in safety set (SS).

#### 4.2 Exposure data

The date, time and dose of drugs given to the subjects should be listed in the statistical analysis report.

#### 4.3 Adverse events

All AE-related information will be provided in the listings of statistical analysis report (including: SAE or not, severity, whether concomitant treatment is given, AE outcome and relationship with study treatment); each AE will be encoded with MedDRA (preferred term (PT), organ system classification (SOC)). The number of AE with different severity and the relationship with study treatment will be summarized by dose group; the incidence and percentage of AE will be summarized and analyzed with preferred term (PT) and organ system classification (SOC) by different dose groups. (AE occurring in all periods is given in the listing, but only TEAE (Treatment Emergent Adverse Events) will be statistically analyzed.)

Double histograms of PK exposure (AUC,  $C_{max}$ ) and AE incidence will be plotted by dose group for naloxone and oxycodone, respectively.

#### 4.3.1 Serious adverse events

Individual SAE data should be listed in the statistical analysis report.

#### 4.4 Evaluation of laboratory tests

For safety set, laboratory examination results of the subjects at the scheduled evaluation point will be summarized by different dose group; meanwhile, the relative changes from the baseline will be summarized by evaluation point. The table for reference (normal) ranges of laboratory parameters will be listed for subjects in each dose group.

The laboratory test results will be classified and summarized by LNH according to lower than (L), equal to (N) or higher than (H) reference range of laboratory parameters.

#### 4.5 Vital signs

All vital sign data will be presented by listing of dose groups and subjects, in which the outliers will be marked. Descriptive statistics and listing of various vital signs and their changes from the baseline after administration will be provided by dose group. For abnormal data, frequency and percentage will be calculated by treatment and abnormality.

#### 4.6 Physical examination

Individual data of physical examination should be listed in statistical analysis report, in which the outliers will be marked. For abnormal data of physical examination, the frequency and percentage will be calculated by treatment and normality.

#### 4.7 ECG evaluation

All ECG data will be listed by dose groups and subjects, while the outliers will be marked. Descriptive statistics of the changes in examination values of ECG parameters relative to baseline after administration will be provided by dose group. For abnormal ECG data, the frequency and percentage will be calculated by dose group and clinical significance.

#### 4.8 Evaluation of pain scores

The pain scores will be summarized at the scheduled evaluation points by different dose groups.

#### 5. Quality control

Statistical analysis and PK analysis should be carried out under the guidance of statisticians and PK experts, and reviewed by relevant quality control personnel.

## 6. List of Tables

## 6.1 List of Tables

| Table 10.1:1 | Trial completion status |
|---|---|
| Table 11.2.1:1 | Demographics results |
| Table 11.3 | Descriptive statistical results of plasma concentrations of oxycodone, naloxone and their metabolites |
| Table 11.4.1.2:1 | Descriptive statistical analysis results (summary) of the PK parameters of oxycodone, |
| | naloxone and their metabolites |
| Table 11.4.1.2:2 | Descriptive statistical analysis results (including individual data) of the PK parameters |
| | of oxycodone, naloxone and their metabolites |
| Table 11.4.1.2:3 | Dose proportionality assessment results |
| Table 12.2.3 | Summary on adverse events |
| Table 12.2.3:1 | Table for severity of adverse events and treatment-related frequency |
| Table 12.2.3:2 | Table for incidence of adverse events (by SOC and PT) |
| Table 12.2.3:3 | Table for frequency analysis of serious adverse events |
| Table 12.4.1:1 | Descriptive statistical analysis results for haematology |
| Table 12.4.1:2 | Descriptive statistical analysis results for changes of haematology relative to the |
| | baseline |
| Table 12.4.1:3 | Table for frequency of haematology results |
| Table 12.4.1:4 | Descriptive statistical analysis results for blood chemistry |
| Table 12.4.1:5 | Descriptive statistical analysis results for changes of haematology relative to the |
| | baseline |
| Table 12.4.1:6 | Table for frequency of blood chemistry results |
| Table 12.4.1:7 | Table for frequency of urinalysis results |
| Table 12.5.1:1 | Descriptive statistical analysis results for vital signs |
| Table 12.5.1:2 | Descriptive statistical analysis results for changes of vital signs relative to the baseline |
| Table 12.5.1:3 | Descriptive statistical analysis results for 12-lead ECG |
| Table 12.5.1:4 | Descriptive statistical analysis results for changes of 12-lead ECG relative to the |
| | baseline |
| Table 12.5.1:5 | Table for frequency of 12-lead ECG results |
| Table 12.5.1:6 | Table for frequency of physical examination results |
| Table 12.5.1:7 | Descriptive statistical analysis results for pain scores |

## 6.2 List of figures

| Figure 1.1 | Mean plasma drug concentration-time linear curve for oxycodone, naloxone and their metabolites |
|---|---|
| Figure 1.2 | Mean plasma drug concentration-time semi-logarithmic curve for oxycodone, naloxone and their metabolites |
| Figure 2.1 | Individual plasma drug concentration-time linear curve for oxycodone, naloxone and |

| | their metabolites |
|---|---|
| Figure 2.2 | Individual plasma drug concentration-time semi-logarithmic curve for oxycodone, |
| | naloxone and their metabolites |

#### 6.3 Table of listings

| Listing11.1.1:1 | Listing of trial completion status |
|-----------------|---------------------------------------------------------|
| Listing11.1.1:2 | Listing of trial protocol deviation |
| Listing11.2.1:1 | Listing of demographics |
| Listing11.3:1 | Listing of Concomitant Medication |
| Listing11.3:2 | Listing of past medical history |
| Listing11.4 | Listing of blood collection |
| Listing12.1:1 | Listing of individual medication |
| Listing12.2.2:1 | Listing of adverse events |
| Listing12.4:1 | Listing of laboratory haematology test results |
| Listing12.4:2 | Listing of laboratory haematology test results |
| Listing12.4:3 | Listing of laboratory blood biochemistry test results |
| Listing12.4:4 | Listing of laboratory blood biochemistry test results |
| Listing12.4:5 | Listing of laboratory urinalysis test results |
| Listing12.5:1 | Listing of individual vital signs results |
| Listing12.5:2 | Listing of individual 12-lead ECG determination results |
| Listing12.5:3 | Listing of individual 12-lead ECG examination results |
| Listing12.5:4 | Listing of individual physical examination results |
| Listing12.5:5 | Listing of individual pain scores results |

## 7. References

- [1] Drug Information Journal, Vol.29, pp. 1039-1048, 1995. Assessment of Dose Proportionality: Report from the Statisticians in the Pharmaceutical Industry/ Pharmacokinetics UK Joint Working Party.
- [2] Brian P. Smith, Francois R. Vandenhende, Karl A. DeSante, Nagy A. Farid, Pamela A. Welch, John T. Callaghan and S. Thomas Forgue. Confidence Interval Criteria for Assessment of Dose Proportionality; Pharmaceutical Research, Vol. 17, No. 10, 2000

## 8. Examples of tables

#### **Tables**

Table 10.1:1 Study completion status

| | TreatmentA | TreatmentB |
|------------------------------------|------------|------------|
| | (N=xx) | (N=xx) |
| | n (%) | n (%) |
| Subjects without taking study drug | XXX | xxx |
| Subjects receiving study drug | xxx | XXX |
| Study completion status | xxx(xx,x) | xxx(xx,x) |
| Withdraw from the trial | | |
| Reason A | xxx(xx,x) | xxx(xx,x) |
| Reason B | xxx(xx,x) | xxx(xx,x) |
| Reason C | xxx(xx,x) | xxx(xx,x) |

N: Number of subjects in each group

Table 10.2.1 Demographics results

| | TreatmentA | TreatmentB |
|------------|--------------|--------------|
| | (N=xx) | (N=xx) |
| Age(years) | | |
| Mean(SD) | xx.x(xx.xx) | xx.x(xx.xx) |
| Median(CV) | xx(xx.xx) | xx(xx.xx) |
| (Min, Max) | (xx,xx) | (xx,xx) |
| Height(cm) | | |
| Mean(SD) | xx.xx(xx.xx) | xx.xx(xx.xx) |

n: Number of subjects with effective data

<sup>%:</sup> N-based percentage

| | TreatmentA | TreatmentB |
|-------------|---------------|---------------|
| | (N=xx) | (N=xx) |
| Median(CV) | xx.xx(xx.xx) | xx.xx(xx.xx) |
| (Min, Max) | (xx.xx,xx.xx) | (xx.xx,xx.xx) |
| Weight(kg) | | |
| Mean(SD) | xx.xx(xx.xx) | xx.xx(xx.xx) |
| Median(CV) | xx.xx(xx.xx) | xx.xx(xx.xx) |
| (Min, Max) | (xx.xx,xx.xx) | (xx.xx,xx.xx) |
| BMI(kg/m^2) | | |
| Mean(SD) | xx.xx(xx.xx) | xx.xx(xx.xx) |
| Median(CV) | xx.xx(xx.xx) | xx.xx(xx.xx) |
| (Min, Max) | (xx.xx,xx.xx) | (xx.xx,xx.xx) |
| Gender | | |
| Male | xx(xx.xx%) | xx.xx(xx.xx) |
| Female | xx(xx.xx%) | xx.xx(xx.xx) |

Table 11.3 Descriptive statistical results of plasma concentrations of oxycodone, naloxone and their metabolites

| | | | | | | | | Sub | ject | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | 1<br>0<br>1 | 1<br>0<br>2 | 1<br>0<br>3 | 1<br>0<br>4 | 1<br>0<br>5 | 1<br>0<br>6 | 1<br>0<br>7 | 1<br>0<br>8 | 1<br>0<br>9 | 1<br>1<br>0 | 1<br>1<br>1 | 1<br>1<br>2 | N | M<br>e<br>a<br>n | S<br>D |
| Tr<br>eat<br>me<br>nt | Analy<br>te | Nomina<br>l_Time<br>(hr) | | | | | | | ( | conc<br>(ng/mL | ) | | | | | | |
| Trea<br>tme<br>nt A | OXN<br>PR | 0.0 | 0.<br>00 | 0.<br>00 | 0.<br>00 | 0.<br>00 | 0.<br>00 | 0.<br>00 | 0.<br>00 | 0.<br>00 | 0.<br>00 | 0.<br>00 | 0.<br>00 | 0.<br>00 | 1 2 | 0.0 | 0.<br>0<br>0 |
| | | 0.5 | 49<br>.6 | 78<br>.6 | 2.<br>19 | 18<br>.3 | 23 | 10<br>.2 | 14<br>9 | 0.<br>60<br>1 | 36<br>.5 | 13<br>.4 | 11<br>1 | 11<br>0 | 1 2 | 67.<br>5 | 7<br>1.<br>2 |
| | | 1.0 | 10<br>8 | 14<br>7 | 64<br>.6 | 24<br>6 | 21<br>7 | 71<br>.2 | 26<br>1 | 40<br>.8 | 12<br>5 | 23<br>7 | 18<br>0 | 18<br>9 | 1 2 | 15<br>7 | 7<br>5.<br>7 |
| | | 1.5 | 14<br>7 | 15<br>1 | 13<br>2 | 17<br>8 | 18<br>9 | 98<br>.8 | 15<br>4 | 10<br>7 | 18<br>7 | 17<br>5 | 14<br>7 | 17<br>6 | 1 2 | 15<br>3 | 2<br>9.<br>7 |
| | | 2.0 | 12<br>5 | 12<br>6 | 14<br>0 | 17<br>5 | 16<br>0 | 11<br>9 | 12<br>4 | 13<br>8 | 19<br>3 | 13<br>3 | 13<br>6 | 14<br>1 | 1 2 | 14<br>2 | 2<br>2.<br>5 |
| | | 3.0 | 12<br>9 | 98<br>.7 | 10<br>6 | 12<br>9 | 11<br>8 | 11<br>4 | 11<br>4 | 84<br>.9 | 14<br>1 | 16<br>5 | 12<br>0 | 12<br>8 | 1 2 | 12<br>1 | 2<br>0.<br>5 |
| | | 4.0 | 13 | .5<br>82 | 87<br>.2 | 10<br>6 | 10<br>6 | 12<br>6 | 10<br>6 | | | 13<br>9 | 89<br>.3 | 10<br>6 | | 10<br>9 | 1<br>7.<br>6 |

Table 11.4.1.2:1 Descriptive statistical analysis results (summary) of the PK parameters of oxycodone, naloxone and their metabolites

| Analyte | Parameters | Units | Treatment A |
|---------|------------------|---------|-------------|
| OXN PR | AUC0_48hr | hr*mg/L | xx(xx) |
| | AUC_%Extrap_pred | % | xx (xx) |
| | AUC0-inf | | xx (xx) |

| Cma | X | ng/mL | xx (xx) |
|-----------|------|-------|------------|
| Tma | X | hr | xx(xx, xx) |
| Lambac | la_z | 1/hr | xx(xx) |
| $T_{1/2}$ | | hr | xx (xx) |

Tmax: Median(Min,Max); Other PK parameters Mean (SD)

Table 11.4.1.2:2 Descriptive statistical analysis results (including individual data) of the PK parameters of oxycodone, naloxone and their metabolites

| Analy<br>te | Treatme<br>nt | statisti<br>cs | Lambada<br>_z<br>(1/hr) | T1/<br>2<br>(hr | Tma<br>x<br>(hr) | Cmax<br>(ng/m<br>L) | AUC0-inf<br>(hr*ng/m<br>L) | %AUCextr<br>ap<br>(%) | AUC0_48<br>hr<br>(hr*mg/L |
|---|---|---|---|---|---|---|---|---|---|
| OXN PR | Treatment A | $\mathbf{N}$ | ** | ** | ** | ** | ** | ** | ** |
| | | Mean | ** | ** | ** | ** | ** | ** | ** |
| | | SD | ** | ** | ** | ** | ** | ** | ** |
| | | Min | ** | ** | ** | ** | ** | ** | ** |
| | | Median | ** | ** | ** | ** | ** | ** | ** |
| | | Max | ** | ** | ** | ** | ** | ** | ** |
| | | CV% | ** | ** | ** | ** | ** | ** | ** |

Table 11.4.1.2:3 Dose proportionality assessment results

| Analyte | Item | Confidence<br>Level | Point<br>Estimate | Confidence<br>Interval | Criterion |
|---|---|---|---|---|---|
| OXN PR | AUC0-48h | 0.1 | xx | (xx, xx) | (0.800,1.250) |
| | AUC0-inf | 0.1 | xx | (xx, xx) | (0.800,1.250) |
| | Cmax | 0.1 | XX | (xx, xx) | (0.800,1.250) |

Table 12.2.3 Summary on adverse events

| Parameter | Treatment A | Treatment B | Total |
|---------------------------------|-------------|-------------|---------|
| | N, N(%) | N, N(%) | N, N(%) |
| All AE | | | |
| Study drug-related AE* | | | |
| Severe AE** | | | |
| Study drug-related severe AE | | | |
| Serious adverse events (SAE) | | | |
| Study drug-related SAE | | | |
| AE leading to study termination | | | |
| AE given combined treatment | | | |
| AE given other treatment | | | |
| AE leading to reduced dose of | | | |
| study drug | | | |

Table 12.2.3:1 Table for severity of adverse events and treatment-related frequency

| Treatment | AE<br>Severity | Definitely<br>related | Probably<br>related | Possibly related | Possibly<br>unrelated | Definitely<br>unrelated | Total |
|---|---|---|---|---|---|---|---|
| TreatmentA (N=12) n (%) | Mild | **(**) | **(**) | **(**) | **(**) | **(**) | |
| | Moderate | **(**) | **(**) | **(**) | **(**) | **(**) | |
| | Severe | **(**) | **(**) | **(**) | **(**) | **(**) | |
| | | 0 0 | • | | | | |

N: Number of subjects in each group

Table 12.2.3:2 Table for incidence of adverse events (by SOC and PT)

| System organ classification<br>GT | | | Treatment B (N=12) |
|---|---|---|---|
| Infection and infectious diseases | Total | **(**) | **(**) |
| | Upper respiratory tract infection | **(**) | **(**) |
| Various types of examinations | Total | **(**) | **(**) |
| | Elevated alanine<br>aminotransferase | **(**) | **(**) |
| | Elevated blood myoglobin | **(**) | **(**) |
| | Elevated creatine<br>phosphokinase | **(**) | **(**) |
| Various types of nervous<br>system diseases | Total | **(**) | **(**) |
| | Head discomfort | **(**) | **(**) |
| Skin and subcutaneous tissue<br>diseases | Total | **(**) | **(**) |
| | Dermatitis | **(**) | **(**) |
| | Rash | **(**) | **(**) |

<sup>\*:</sup> Positively related, probably related and possibly related are regarded to be correlated with the study drug

<sup>\*\*:</sup> The severity of AE is SAE

N, N(%): Nbr of AE, Nbr of Subject(incidence)

n: Number of subjects with effective data

<sup>%:</sup> N-based percentage

| System organ classification GT | Standard name of AE<br>PT | Treatment A (N=12) | Treatment B (N=12) |
|---|---|---|---|
| Systemic disease and various administration site reactions | Total | **(**) | **(**) |
| | Fatigue | **(**) | **(**) |
| | Local reaction | **(**) | **(**) |
| | Drowsiness | **(**) | **(**) |
| Kidneys and urinary system diseases | Total | **(**) | **(**) |
| | Frequent micturition | **(**) | **(**) |
| Gastrointestinal diseases | Total | **(**) | **(**) |
| | Constipation | **(**) | **(**) |
| | Abdominal pain | **(**) | **(**) |
| | Diarrhea | **(**) | **(**) |
| | Oral ulcer | **(**) | **(**) |
| Blood and lymphatic system<br>diseases | Total | **(**) | **(**) |
| | Neutropenia | **(**) | **(**) |
| Eye diseases | Total | **(**) | **(**) |
| | Conjunctival hyperemia | **(**) | **(**) |

Table 12.2.3:3 Table for frequency analysis of serious adverse events

| | SAE related to | |
|------------------|----------------|--------|
| Treatment | study drug(%) | SAE(%) |
| ** | ** | ** |
| * Absence of SAE | | |

Table 12.4.1:1 Descriptive statistical analysis results for haematology

| Treatment | Item | Unit | ExpDelta (min) | N | Mean | SD | CV(%) | Min | Median | Max |
|---|---|---|---|---|---|---|---|---|---|---|
| Treatment A | Item1 | U/L | TimePoint1 | ** | ** | ** | ** | ** | ** | ** |
| | | | TimePoint2 | ** | ** | ** | ** | ** | ** | ** |
| | | | | ** | ** | ** | ** | ** | ** | ** |
| | Item2 | U/L | TimePoint1 | ** | ** | ** | ** | ** | ** | ** |

| Treatment | Item | Unit | ExpDelta (min) | N | Mean | SD | CV(%) | Min | Median | Max |
|---|---|---|---|---|---|---|---|---|---|---|
| · | | · | TimePoint2 | ** | ** | ** | ** | ** | ** | ** |
| | | | | ** | ** | ** | ** | ** | ** | ** |
| | Item3 | g/L | TimePoint1 | ** | ** | ** | ** | ** | ** | ** |
| | | | TimePoint2 | ** | ** | ** | ** | ** | ** | ** |
| | | | | ** | ** | ** | ** | ** | ** | ** |
| | Item4 | mmol/L | TimePoint1 | ** | ** | ** | ** | ** | ** | ** |
| | | | TimePoint2 | ** | ** | ** | ** | ** | ** | ** |
| | | | | ** | ** | ** | ** | ** | ** | ** |

Screening:TimePoint\*\*—TimePoint\*\*;Baseline:TimePoint\*\*—TimePoint\*\*;Treatment:TimePoint\*\*—TimePoint\*\*;

Similar tables are as follows

Table 12.4.1:2 Descriptive statistical analysis results for changes of haematology relative to the baseline

Table 12.4.1:4 Descriptive statistical analysis results for blood chemistry

Table 12.4.1:5 Descriptive statistical analysis results for changes of haematology relative to the baseline

Table 12.5.1:1 Descriptive statistical analysis results for vital signs

Table 12.5.1:2 Descriptive statistical analysis results for changes of vital signs relative to the baseline

Table 12.5.1:3 Descriptive statistical analysis results for 12-lead ECG

Table 12.5.1:4 Descriptive statistical analysis results for changes of 12-lead ECG relative to the baseline

Table 12.4.1:3 Table for frequency of haematology results

| Treatment | Item | ExpDelta<br>(min) | Norma l n(%) | Abnormal, without clinical significance n(%) | Abnormal, with clinical significance n(%) |
|---|---|---|---|---|---|
| Treatment A | Item<br>1 | TimePoint | **(**) | **(**) | **(**) |
| | | TimePoint 2 | **(**) | **(**) | **(**) |
| | | | **(**) | **(**) | **(**) |
| | Item 2 | TimePoint | **(**) | **(**) | **(**) |
| | | TimePoint 2 | **(**) | **(**) | **(**) |
| | | | **(**) | **(**) | **(**) |

| Treatment | Item | ExpDelta<br>(min) | Norma<br>l<br>n(%) | Abnormal, without clinical significance n(%) | Abnormal, with clinical<br>significance<br>n(%) |
|---|---|---|---|---|---|
| | Item 3 | TimePoint | **(**) | **(**) | **(**) |
| | | TimePoint 2 | **(**) | **(**) | **(**) |
| | | | **(**) | **(**) | **(**) |
| | Item<br>4 | TimePoint | **(**) | **(**) | **(**) |
| | | TimePoint 2 | **(**) | **(**) | **(**) |
| | | | **(**) | **(**) | **(**) |

Screening: TimePoint\*\*--TimePoint\*\*; Baseline: TimePoint\*\*--TimePoint\*\*; Treatment: TimePoint\*\*---TimePoint\*\*.

#### Similar tables are as follows

Table 12.4.1:6 Table for frequency of blood chemistry results

Table 12.4.1:7 Table for frequency of urinalysis results

Table 12.5.1:5 Table for frequency of 12-lead ECG results

Table 12.5.1:6 Table for frequency of physical examination results

#### **Figures**

Figure 1.1 Mean plasma drug concentration-time linear curve for oxycodone, naloxone and their metabolites



Similar figures are as follows

Figure 1.2 Mean plasma drug concentration-time semi-logarithmic curve for oxycodone, naloxone and their metabolites

Figure 2.1 Individual plasma drug concentration-time linear curves for oxycodone, naloxone and their metabolites



Similar figures are as follows,

Figure 2.2 Individual plasma drug concentration-time semi-logarithmic curve for oxycodone, naloxone and their metabolites

## Listing

Listing11.1.1:1 listing of trial completion status

| Subject | Treatment | Completion<br>status | Completion<br>date | Signature of<br>Investigator<br>(Date) |
|---|---|---|---|---|
| 1001 | Treatment A | ** | ** | ** |
| 1002 | Treatment A | ** | ** | ** |
| 1003 | Treatment A | ** | ** | ** |
| 1004 | Treatment A | ** | ** | ** |

Listing 11.1.1:2 Listing of trial protocol deviation

| Treatment | Occasion | Subject | (PI<br>endorsed)<br>measures<br>taken on<br>protocol<br>deviation | Actual situation of deviation events | Nature<br>of<br>protocol<br>deviation | Time of protocol deviation | Protocol<br>requirements<br>for deviation<br>event-related<br>items |
|---|---|---|---|---|---|---|---|
| ** | ** | ** | ** | ** | ** | ** | ** |
| | | ** | ** | ** | ** | ** | ** |

Listing 11.2.1:1 Listing of demographics

| | | | | <u> </u> | | |
|---------|---------|-----|------|----------|------|----------|
| | | | | Heig | Weit | |
| | Age | Gen | | ht | ht | BMI |
| Subject | (Years) | der | Race | (m) | (kg) | (kg/m^2) |
| ** | ** | ** | ** | ** | ** | ** |
| ** | ** | ** | ** | ** | ** | ** |
| | | | ••• | | | |

Listing11.3:1 Listing of Concomitant Medication

| Treat<br>nt | | Occasio<br>n | Subje<br>ct | Does concomita nt medicatio n or treatment occur before the first dose? | Dru<br>g<br>nam<br>e | Dos<br>e<br>unit | Indicatio<br>n | Dosage for<br>single-dose<br>administrati<br>on | Route of<br>administrati<br>on | Does medicatio n continue at ending of this study? | Dosing<br>frequen | Startin<br>g time | Endin<br>g time |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| ** | : | ** | ** | ** | ** | ** | ** | ** | ** | ** | ** | ** | ** |
| ** | | ** | ** | ** | ** | ** | ** | ** | ** | ** | ** | ** | ** |
| ** | : | ** | ** | ** | ** | ** | ** | ** | ** | ** | ** | ** | ** |

Listing 11.3:2 Listing of past medical history

| | Preferred | | |
|---------|------------|---------------------------------|-------|
| Subject | Term | PT annotations | Value |
| ** | Admissions | Past history of hospitalization | ** |
| | Operations | Past history of surgery/trauma | ** |
| | ** | ** | ** |

| P | referred | | |
|---------|-----------|---------------------------------|-------|
| 'ubject | Term | PT annotations | Value |
| | ** | ** | ** |
| | ** | ** | ** |
| | ** | ** | ** |
| | ** | ** | ** |
| | ** | ** | ** |
| | ** | ** | ** |
| | ** | ** | ** |
| 1002 Ad | lmissions | Past history of hospitalization | ** |
| Op | perations | Past history of surgery/trauma | ** |
| | ** | ** | ** |
| | ** | ** | ** |

Listing 11.4 Listing of blood collection

| Subject | Treatment | Expected<br>delta-time<br>(hr) | Actual<br>Time<br>(hr) | BiasTime<br>(hr) | Flag | status |
|---|---|---|---|---|---|---|
| ** | ** | 0 | ** | ** | ** | ** |
| | | 0.5 | ** | ** | ** | ** |
| | | 1 | ** | ** | ** | ** |
| | | 1.5 | ** | ** | ** | ** |
| | | 2 | ** | ** | ** | ** |
| | ** | 0 | ** | ** | ** | ** |
| | | 0.5 | ** | ** | ** | ** |
| | | 1 | ** | ** | ** | ** |
| | | 1.5 | ** | ** | ** | ** |
| | | 2 | ** | ** | ** | ** |

Listing 12.1:1 Listing of individual medication

| Subject | Occasion | Treatment | Expected time (min) | Actual delta time (min) | Admin time (Day and<br>Time) |
|---|---|---|---|---|---|
| ** | ** | ** | ** | ** | ** |
| ** | ** | ** | ** | ** | ** |
| ** | ** | ** | ** | ** | ** |
| ** | ** | ** | ** | ** | ** |
| ** | ** | ** | ** | ** | ** |

Listing 12.2.2:1 Listing of adverse events

| | | | | ~ | | AE | AE | | Relationship |
|---|---|---|---|---|---|---|---|---|---|
| | | | | System organ | AE | beginning | ending | Whether | between AE and |
| Treatment | Occasion | SubjectNr | PT | | severity | time | time | SAE | treatment |
| ** | ** | ** | ** | ** | ** | ** | ** | ** | ** |
| ** | ** | ** | ** | ** | ** | ** | ** | ** | ** |
| ** | ** | ** | ** | ** | ** | ** | ** | ** | ** |
| ** | ** | ** | ** | ** | ** | ** | ** | ** | ** |

Listing 12.4:1 Listing of laboratory haematology test results

| Subject | Treatment | | Time<br>(min) | Item | Value | Notes |
|---------|-----------|----|---------------|-------------|-------|-------|
| ** | ** | ** | ** | LabHae<br>m | ** | ** |
| | ** | ** | ** | LabHae<br>m | ** | ** |
| | ** | ** | ** | LabHae<br>m | ** | ** |
| | ** | ** | ** | LabHae<br>m | ** | ** |

| Subject | Treatment | Occasion | (min) | Item | Value | Note. |
|---------|-----------|----------|-------|------|-------|-------|
|---------|-----------|----------|-------|------|-------|-------|

Similar listings are as follows,

Listing 12.4:3 Listing of laboratory blood biochemistry test results

Listing 12.4:5 Listing of laboratory urinalysis test results

Listing 12.5:2 Listing of individual 12-lead ECG determination results

Listing 12.5:4 Listing of individual physical examination results

Listing 12.4:2 Listing of laboratory haematology test results

| | | | Time | | | | Lower | Upper | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Subject | Treatment | Occasion | (min) | Item | Unit | Value | Limit | Limit | Notes | Judge |
| ** | ** | ** | ** | Item1 | ** | ** | ** | ** | ** | ** |
| | | | | Item2 | ** | ** | ** | ** | ** | ** |
| | | | | Item3 | ** | ** | ** | ** | ** | ** |

Similar listings are as follows,

Listing 12.4:4 Listing of laboratory blood biochemistry examination results

Listing 12.5:1 Listing of individual vital signs results

Listing 12.5:3 Listing of individual 12-lead ECG examination results